CLINICAL TRIAL: NCT02585557
Title: Heart Health NOW (Previously Known as Facilitation, Spread, and Translation of Patient-Centered Evidence in North Carolina Practices)
Brief Title: Heart Health NOW (Previously Known as FAST PACE NC)
Acronym: HHN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-0479; 1R18HS023912-01 (AHRQ)
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cluster A (Experimental): 50 practices randomly assigned to start intervention at month 9. Assigned Intervention: Primary Care Practice Support. The intervention consists of practice facilitation, academic detailing, and regional learning collaboratives.
  Interventions: Other: Primary Care Practice Support
- Cluster B (Experimental): 50 practices randomly assigned to start intervention at month 11. Assigned Intervention: Primary Care Practice Support. The intervention consists of practice facilitation, academic detailing, and regional learning collaboratives.
  Interventions: Other: Primary Care Practice Support
- Cluster C (Experimental): 50 practices randomly assigned to start intervention at month 12. Assigned Intervention: Primary Care Practice Support. The intervention consists of practice facilitation, academic detailing, and regional learning collaboratives.
  Interventions: Other: Primary Care Practice Support
- Cluster D (Experimental): 50 practices randomly assigned to start intervention at month 14. Assigned Intervention: Primary Care Practice Support. The intervention consists of practice facilitation, academic detailing, and regional learning collaboratives.
  Interventions: Other: Primary Care Practice Support
- Cluster E (Experimental): 50 practices randomly assigned to start intervention at month 16. Assigned Intervention: Primary Care Practice Support. The intervention consists of practice facilitation, academic detailing, and regional learning collaboratives.
  Interventions: Other: Primary Care Practice Support

INTERVENTIONS:
Other: Primary Care Practice Support — The intervention consists of practice facilitation, academic detailing, and regional learning collaboratives.

SUMMARY:
The objective of this study is to determine if primary care practice support accelerates the dissemination and implementation of patient-centered outcome results (PCOR) findings to improve heart health and increases primary care practices' capacity to incorporate other PCOR findings in the future.

DETAILED DESCRIPTION:
The burden of cardiovascular disease in North Carolina remains large. The latest data available show an annual cardiovascular death rate of 263 per 100,000 explaining almost one-third of deaths in the state. Disease progression is largely determined by several risk factors including elevated blood pressure or cholesterol, not using aspirin for prevention, and tobacco use. Primary care practices as currently organized have been unable to get more than half these patients to achieve recommended targets for risk factor reduction. Small independent practices, in particular, lack resources for enhanced practice support to improve cardiovascular care.

This study will enroll 300 primary care practices to evaluate the effect of primary care support on evidence-based cardiovascular disease (CVD) prevention and organizational change process measures. Each practice will start the trial as a control, receive the intervention at a randomized time point, and then enter a maintenance period 12 months after starting the intervention. All practices will receive 12 months of the intense intervention including onsite quality improvement (QI) facilitation, academic detailing, electronic health record (EHR) support, and, through the North Carolina Health Information Exchange (HIE), a shared statewide utility providing whole population analytics, care gap identification, benchmarking, and an external reporting mechanism which otherwise would not be available to independent practices.

A successful intervention would prove that practice facilitation supported by effective informatics tools is an effective method of translating PCOR findings into practice. Discernible reductions in cardiovascular risk in 300 practices covering over an estimated 900,000 adult patients would likely lead to prevention of thousands of cardiovascular events within 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Primary care practice in North Carolina with 10 or fewer providers in a single location
* must have implemented an EHR and either be connected to or have agreed to connect to the HIE.

Exclusion Criteria:

* practices with more than 10 providers in a single location
* practices receiving practice facilitation services beyond the usual support provided by Area Health Education Centers (AHEC) or the Community Care of North Carolina (CCNC) program through their parent organization.
* practices without an EHR
* practices where the central practice organization either bars the practice from our program or provides onsite facilitation services equal to or greater than the 4-6 hour standard contact with a QI coach

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Measurable reduction in arteriosclerotic cardiovascular disease (ASCVD) risk | 18 months
  By comparing EHR data at baseline and post-intervention, determine whether practice support resulted in discernible reduction in CVD risk.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Cykert, MD, Principal Investigator — UNC Chapel Hill

IPD SHARING:
Plan to Share IPD: No
Will share data on practice improvement. Practices receive data relevant to reducing their patients cardiovascular risk. The practice then receives advice on practice redesign and population management to improve, standard, clinical, chronic care measures. There is no experimental, direct patient intervention.

REFERENCES:
- [Derived] Weiner BJ, Pignone MP, DuBard CA, Lefebvre A, Suttie JL, Freburger JK, Cykert S. Advancing heart health in North Carolina primary care: the Heart Health NOW study protocol. Implement Sci. 2015 Nov 14;10:160. doi: 10.1186/s13012-015-0348-4. PMID 26577091